CLINICAL TRIAL: NCT05301491
Title: Investigation of the Effects of Dance Therapy on Balance, Falling, Body Awareness and Functionality in Women With Chronic Low Back Pain
Brief Title: The Effects of Dance Therapy in Women With Chronic Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hasan Kalyoncu University (Other)
Responsible Party: Principal Investigator, Elif Dinler, Research assistant, Hasan Kalyoncu University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021/025
Record Dates: First submitted 2022-02-25; First posted 2022-03-29 (Actual); Last update posted 2022-08-11 (Actual); Status verified 2022-08

CONDITIONS: Low Back Pain; Chronic Pain; Chronic Low-back Pain
Keywords: Low back pain; Chronic low back pain; Dance Therapy; Balance; Falling risk; Functionality; Body awareness
MeSH Terms: conditions — Low Back Pain; Chronic Pain | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Two randomized controlled groups
  Forty female patients who were diagnosed with chronic low back pain and met the inclusion criteria of the study were divided into two groups.These individuals are going to be divided into groups as the odd numbers to study group and even numbers to the control group.
  Inclusion criteria of patients;
  * Those who agree to participate in the study voluntarily
  * Having low back pain lasting longer than 3 months,
  * Having values between 4 and 7 on the Visual Analog Scale.
  * Female individuals between the ages of 18-65
  Exclusion criteria of patients; Those with a Body Mass Index (BMI) greater than 35 kg/m², pregnant women, those with following problems; neural findings, malignancy, inflammation, arthritis, metabolic bone disease, column vertebralis or lower extremity surgery, cardiovascular system diseases, severe osteoporosis, communication and hearing disorders, and those who illiterate, receive other treatment for low back pain.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dance therapy group (Experimental): This group included in the dance therapy program throughout the study.
  Interventions: Other: Dance Therapy Group; Other: Pyhsiotherapy Modalities
- Control group (Experimental): This group included in the conventional low back pain exercise program throughout the study.
  Interventions: Other: Exercise Group; Other: Pyhsiotherapy Modalities

INTERVENTIONS:
Other: Dance Therapy Group — Dance therapy group patients are going to be treated 3 days a week for 8 weeks. Patients who started treatment are going to be randomly divided into groups that includes four individuals, due to COVID-19 pandemic preventions.
  Dance therapy is going to be applied with individualized choreographies specially prepared for the patients, taking the expert opinion of the dance therapist. Choreographies of different dance genres (step/aerobic dance, zumba, salsa, bachata, oriental etc.) are going to be used in the program. Sessions are going to be with the practitioner in a bright, clean, empty and noiseless room in front of a full-length wall mirror. The practitioner is going to participate to dance therapy throughout the sessions, allowing patients to imitate movements. Session duration is going to be 40 minutes. Patients will be given a one-minute rest period during music transitions.
  Other Names: Study Group
  Arms: Dance therapy group
Other: Exercise Group — The patients in the control group is going to perform conventional low back exercises. The program of the patients will start with stretching and warming exercises, and will continue with strengthening exercises.
  Exercises planed for control group;
  1. Unilateral hip-knee flexion (self-assisted exercise)
  2. Bilateral hip-knee flexion (self-assisted exercise)
  3. Straight leg lifting with the aid of a sheet/rigid band
  4. Posterior pelvic tilt
  5. Bridge building exercise
  6. Cat-camel exercise
  7. Half shuttle in sagittal plane
  8. Right and left rotational shuttle
  9. Trunk hyperextension in prone position
  10. Rotational exercise with hip-knee flexed in supine position Patients are going to do exercises with ten repetitions. As the sessions progressed, the number of repetitions will be increased.
  Other Names: Control Group
  Arms: Control group
Other: Pyhsiotherapy Modalities — 20 minutes hotpack, 3-5 minutes ultrasound and 20 minutes conventional type Transcutaneous Electrical Nerve Stimulation (TENS) are going to be applied to lumbar region of all patients in prone position.
  Other Names: Both Groups

SUMMARY:
The aim of this study is to investigate the effect of dance therapy on balance, falling, body awareness and functionality parameters in patients with chronic low back pain. As a result of our study, it is thought that dance therapy will positively affect balance, falling, body awareness and functionality in patients with chronic low back pain compared to conventional therapy.

H 1: Dance therapy improves balance in women with chronic low back pain.

H 2: Dance therapy reduces the risk of falling in women with chronic low back pain.

H 3: Dance therapy increases body awareness in women with chronic low back pain.

H 4: Dance therapy increases functionality in women with chronic low back pain.

H 5: Dance therapy provides more improvement in the parameters investigated compared to conventional therapy in women with chronic low back pain.

DETAILED DESCRIPTION:
Individuals diagnosed with chronic low back pain and meeting the inclusion criteria are going to be included in the study. These individuals are going to be divided into groups as the odd numbers to study group and even numbers to the control group. Hotpack, ultrasound and Transcutaneous Electrical Nerve Stimulation (TENS) are going to be applied to the patients in the both groups for 3 days a week for 2 months. Besides that, control group is going to perform 40-minute classical exercise program 3 days a week for 2 months. Study group is going to perform dance therapy protocol as indicated below;

* 10 minutes warm-up (stepping),
* 25 minutes of dance (such as; steps, figures using hip and knee flexions, hip circulation, and hip rotations)
* 5 minutes stretching (relaxation) exercises.

Demographic information form is going be filled out patients including information about; age, height (cm), weight (kg), occupation, educational status, bilateral leg length (cm), previous and present diseases, waist/hip ratio, previous surgeries, trunk range of motions, low back pain duration, smoking, falling story. Additionally, following questionnaires are going to be applied to both groups;

* Short Form Mc Gill Pain Questionnaire,
* Oswestry Disability Index,
* Body Awareness Ratio Questionnaire,
* Nottingham Health Profile Questionnaire,
* Tampa Kinesiophobia Scale,
* The World Health Organization Quality of Life (WHOQoL) Scale,
* Y balance test
* Time Up and Go (TUG) test

SPSS version 23 (SPSS Inc, Armonk, NY) program will be used in the analysis of the data. Mann Whitney U test, Wilcoxon test and student t test will be analyse methods.

ELIGIBILITY:
Inclusion criteria;

* Those who agree to participate in the study voluntarily
* Having low back pain lasting longer than 3 months,
* Having values between 4 and 7 on the Visual Analog Scale.
* Female individuals between the ages of 18-65

Exclusion criteria; Those with a Body Mass Index (BMI) greater than 35 kg/m², pregnant women, those with following problems; neural findings, malignancy, inflammation, arthritis, metabolic bone disease, column vertebralis or lower extremity surgery, cardiovascular system diseases, severe osteoporosis, communication and hearing disorders, and those who illiterate, receive other treatment for low back pain.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — The study is going to be conducted only with female patients.
Enrollment: 40 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-05-30 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Y balance test score | 8 weeks
  Balance score is going to be assess by Y balance test to determine change from baseline.
Change from baseline in Time Up and Go test seconds | 8 weeks
  Falling risk is going to be assess by Time Up and Go test seconds to determine change from baseline.
Change from baseline in body awareness ratio score | 8 weeks
  Body awareness ratio score is going to be assess by Body Awareness Ratio Questionnaire to determine change from baseline.
Change from baseline in functionality score | 8 weeks
  Functionality score is going to be assess by Oswestry Disability Index to determine change from baseline.

SECONDARY OUTCOMES:
Change from baseline in range of motion degree | 8 weeks
  Range of motion degree is going to be assess by goniometric measurement to determine change from baseline.
Change from baseline in waist/hip ratio | 8 weeks
  Waist/hip ratio is going to be assess by measuring tape from waist and hip circumference to determine change from baseline.
Change From Baseline in Pain Scores | 8 weeks
  Pain score is going to be assess by Short Form Mc Gill Pain Questionnaire to determine change from baseline.
Change from baseline in kinesiophobia score | 8 weeks
  Kinesiophobia score is going to be assess by Tampa Kinesiophobia Scale to determine change from baseline.
Change from baseline in quality of life score | 8 weeks
  Quality of life score is going to be assess by WHOQoL Questionnaire to determine change from baseline.
Change from baseline in perceived health status score | 8 weeks
  Perceived health status score is going to be assess by Nottingham Health Profile Questionnaire to determine change from baseline.

CONTACTS AND LOCATIONS:
Locations (1):
- Hasan Kalyoncu University, Gaziantep, Turkey (Türkiye)